CLINICAL TRIAL: NCT05527223
Title: Integrated Care with GP Participation for Older Persons in the Ambulatory Care Hub: a Prospective Cohort Study of Clinical and Process Outcomes.
Brief Title: Integrated Care with GP Participation for Older Persons in the Ambulatory Care Hub: a Prospective Cohort Study.
Status: Completed | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: 116/2021
Record Dates: First submitted 2022-08-11; First posted 2022-09-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Comprehensive Geriatric Assessment
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Comprehensive Geriatric Assessment (CGA) demonstrates positive outcomes amoung community-dwelling older people living with frailty. However, there is currently no evidence of benefit for CGA with General Practitioner (GP) participation within the Irish Primary Care setting. This study aims to explore the clinical and process outcomes of older adults living with frailty who are screened by and referred to one of the three Ambulatory Care Hub's in the primary care setting in the Mid-West of Ireland by their GP, where they undergo a CGA .

DETAILED DESCRIPTION:
The growth of ageing population poses significant difficulties in the delivery of healthcare to older adults. As people age, they experience a decline in their intrinsic capacities which leads to an increasing prevalence of multi-morbidity which ultimately leads to older adults at increased risk of requiring emergency care and increased multidisciplinary health needs.

With functional decline and deterioration in an older persons' ability to self-care being a common consequence of hospitalisation, older people are placed at higher risk of requiring increased care needs after discharge from acute care and transfer between care settings proves a challenge for the provision of seamless quality care.

The World Health Organisation recommends health and social care professionals intervening at an early stage of this ageing process in order to prevent or delay the process of becoming frail through delivering effective interventions that are targeted at functional decline. Internationally, there is recognition for health and social care systems to reorient towards longitudinal, preventive, coordinated and integrated care models, reflecting the growth in multi-morbidity and the needs of older people's complex health and social care requirements. The World Health Organisation acknowledges this shift in healthcare delivery and launched the 'WHO Guidelines on Integrated Care for Older People' programme where it highlighted the need to develop and implement comprehensive community-based approaches at the primary healthcare level in the context of a needs assessment and integrated care plan.

CGA is an interdisciplinary diagnostic process which includes an assessment and holistic management plan that is based on the individual needs of the older person. As many older adults' first point of contact with the health service is through primary care, General Practitioners (GPs) play a crucial role in the coordination of the older person's care.

Frailty screening by the GP and comprehensive geriatric assessment within the primary care setting has demonstrated significant positive health outcomes in community-dwelling older people, demonstrating reduced rates of hospitalisation, reduced hospital re-admissions, reduced GP visits and an increase in social activities.

A primary care based multidisciplinary team aim to improve the delivery of care and clinical and process outcomes for community-dwelling older people through the delivery of CGA in the Ambulatory Care Hub (ACH). An ACH is a clinical site within the primary care setting, with access to diagnostics, specialised services and specialist care in order to support older people to live in their own homes for as long as possible.

This study aims to explore the clinical and process outcomes of older adults living with frailty who are screened by and referred to one of the three Ambulatory Care Hub's in the Mid-West of Ireland by their GP.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the ACH by their GP
* Score between 4 and 6 on the Rockwood Clinical Frailty Scale
* Reside within CHO 3 and the catchment area of the relevant ACH hub
* Have been assessed in-person by the referrer
* Has not had MDT input within the last three months

And any one of the following criteria:

* Fall within the last month unrelated to acute cardiac or neurological cause & no previous falls assessment
* Increased dependency or increased carer burden in the last month
* A deterioration in swallow in the last month including symptoms of recurrent chest infections
* Weight loss
* Coughing when eating/drinking
* Self-modifying diet secondary to difficulties or experienced an adverse drug reaction within the last month excluding allergic reaction.

Exclusion Criteria:

Patients will be excluded if they:

* Present with an acute neurological or cardiovascular event
* Are more appropriate to an alternative care pathway or service e.g. primary care or geriatric medicine clinic
* Present with injuries, unless the injury has already been appropriately managed,
* Are experiencing an acute medical illness requiring treatment in an acute hospital setting
* If care is being provided by other health care professionals at the time of referral and it is apparent that they are working to meet goals aligned with the current service
* They require investigation or treatment not available in the relevant ICPOP hub (unless these investigations are already being arranged elsewhere)
* They have had MDT input in the last three months
* Have confirmed or suspected Covid-19 infection
* Or other exclusions at the discretion of the integrated care team based on clinical expertise and available resource.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All older adults aged ≥75 years who are referred to the ACH by their GP between February 2022 and January 2023 (inclusive) will be considered eligible for participation in the study, if they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of functional decline | 30-days
  The number of participants who experience functional decline or do not as measured by the Barthel Index (BI). Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported BI. The sum of all of the 10 subscales of the BI ranges from 0-20 points where a higher score indicates increased independence.
Incidence of functional decline | 6-months
  The number of participants who experience functional decline or do not as measured by the Barthel Index (BI). Functional decline is defined as a net decrease in the number of activities of daily living performed independently as measured by the self-reported BI. The sum of all of the 10 subscales of the BI ranges from 0-20 points where a higher score indicates increased independence.

SECONDARY OUTCOMES:
Primary healthcare use (within and outside of ACH healthcare utilisation) | 30-days
  Number of services that participants were in receipt of following index visit at the ACH including; GP visits, Public Health Nurse visits, Health and Social Care Professional use, formal homecare support. This will be categorised by healthcare use linked to the ACH and outside of the ACH.
Primary healthcare use (within and outside of ACH healthcare utilisation) | 6-months
  Number of services that participants were in receipt of following index visit at the ACH including; GP visits, Public Health Nurse visits, Health and Social Care Professional use, formal homecare support. This will be categorised by healthcare use linked to the ACH and outside of the ACH.
Secondary healthcare use | 30-days
  Number of secondary healthcare services that participants were in receipt of including; Outpatient services, ED presentation and unplanned hospital admission.
Secondary healthcare use | 6-months
  Number of secondary healthcare services that participants were in receipt of including; Outpatient services, ED presentation and unplanned hospital admission.
Quality of integrated care from the perspective of participants | 30-days
  Participants evaluate the quality of integrated care across a number of domains using the Patient Assessment of Integrated Elderly Care Questionnaire. The sum of all subscales may range from 0-100, where a higher score reflects better perceived quality of care.
Health related quality of life (HRQOL) | 30-days
  Participants will rate their HRQOL using the EuroQoL-5D-5L where the sum of 5 subscales may range from 5-25 where 5 points indicates the lowest possible HRQOL and 25 indicates the highest. The participant must also rate their health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' on a scale of 0-100.
Health related quality of life (HRQOL) | 6-months
  Participants will rate their HRQOL using the EuroQoL-5D-5L where the sum of 5 subscales may range from 5-25 where 5 points indicates the lowest possible HRQOL and 25 indicates the highest. The participant must also rate their health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' on a scale of 0-100.
Mortality | 30-days
  The number of participants who died following their index visit at the ACH
Mortality | 6-months
  The number of participants who died following their index visit at the ACH
Nursing home admission | 30-days
  Number of participants who were admitted to a nursing home or residential care facility following their index visit to the ACH
Nursing home admission | 6-months
  Number of participants who were admitted to a nursing home or residential care facility following their index visit to the ACH

CONTACTS AND LOCATIONS:
Overall Officials: Rose Galvin, Study Director — University of Limerick
Locations (1):
- School of Allied Health, University of Limerick., Limerick, Munster, Ireland

REFERENCES:
- [Background] Liljas AEM, Brattstrom F, Burstrom B, Schon P, Agerholm J. Impact of Integrated Care on Patient-Related Outcomes Among Older People - A Systematic Review. Int J Integr Care. 2019 Jul 24;19(3):6. doi: 10.5334/ijic.4632. PMID 31367205
- [Background] Mann J, Thompson F, McDermott R, Esterman A, Strivens E. Impact of an integrated community-based model of care for older people with complex conditions on hospital emergency presentations and admissions: a step-wedged cluster randomized trial. BMC Health Serv Res. 2021 Jul 16;21(1):701. doi: 10.1186/s12913-021-06668-x. PMID 34271945
- [Background] World Health Organisation. Integrated Care for older people: Realigning primary health care to respond to population ageing. 2018.
- [Background] Everink IHJ, van Haastregt JCM, Tan FES, Schols JMGA, Kempen GIJM. The effectiveness of an integrated care pathway in geriatric rehabilitation among older patients with complex health problems and their informal caregivers: a prospective cohort study. BMC Geriatr. 2018 Nov 16;18(1):285. doi: 10.1186/s12877-018-0971-4. PMID 30445923
- [Background] Roe L, Normand C, Wren MA, Browne J, O'Halloran AM. The impact of frailty on healthcare utilisation in Ireland: evidence from the Irish longitudinal study on ageing. BMC Geriatr. 2017 Sep 5;17(1):203. doi: 10.1186/s12877-017-0579-0. PMID 28874140
- [Background] Briggs R, McDonough A, Ellis G, Bennett K, O'Neill D, Robinson D. Comprehensive Geriatric Assessment for community-dwelling, high-risk, frail, older people. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012705. doi: 10.1002/14651858.CD012705.pub2. PMID 35521829
- [Background] Glynn LG, Valderas JM, Healy P, Burke E, Newell J, Gillespie P, Murphy AW. The prevalence of multimorbidity in primary care and its effect on health care utilization and cost. Fam Pract. 2011 Oct;28(5):516-23. doi: 10.1093/fampra/cmr013. Epub 2011 Mar 24. PMID 21436204
- [Background] World Health Organization. World report on ageing and health: World Health Organization; 2015
- [Derived] Hayes C, Whiston A, Fitzgerald C, Devlin C, Condon B, Manning M, Leahy A, Robinson K, Galvin R. Community Specialist Teams for Older Persons (CST-OP) at risk of, or living with frailty in Ireland: a prospective cohort study of a new model of integrated care for community dwelling older adults. BMC Prim Care. 2025 Jun 5;26(1):193. doi: 10.1186/s12875-025-02895-x. PMID 40474059